CLINICAL TRIAL: NCT04074356
Title: Non-invasive Markers of Esophageal Function in Adults
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Vanderbilt University Medical Center (Other)
Responsible Party: Principal Investigator, Dhyanesh Patel, Principal Investigator, Vanderbilt University Medical Center
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 191280
Record Dates: First submitted 2019-08-28; First posted 2019-08-30 (Actual); Last update posted 2025-09-05 (Actual); Status verified 2025-08

CONDITIONS: Dysphagia
MeSH Terms: conditions — Deglutition Disorders

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (3):
- Healthy Controls (Active Comparator): Healthy volunteers with no known gastrointestinal complications will be given questionnaires and testing by electroesophagogram (EESG) and magnetoesophagogram (MESG).
  Interventions: Other: Clinical measure questionnaires; Diagnostic Test: EESG; Diagnostic Test: MESG
- Achalasia subjects (Active Comparator): Subjects who have undergone standard of care high resolution manometry that results in a diagnosis of achalasia will be given questionnaires and testing by electroesophagogram (EESG) and magnetoesophagogram (MESG).
  Interventions: Other: Clinical measure questionnaires; Diagnostic Test: EESG; Diagnostic Test: MESG; Diagnostic Test: High resolution manometry (HRM)
- Hypercontractile/spastic disorder subjects (Active Comparator): Subjects who have undergone standard of care high resolution manometry that results in a diagnosis of hypercontractile/spastic disorder will be given questionnaires and testing by electroesophagogram (EESG) and magnetoesophagogram (MESG).
  Interventions: Other: Clinical measure questionnaires; Diagnostic Test: EESG; Diagnostic Test: MESG; Diagnostic Test: High resolution manometry (HRM)

INTERVENTIONS:
Other: Clinical measure questionnaires — Collection of patient reported symptoms and perception of health
Diagnostic Test: EESG — Use of silver-silver chloride cutaneous electrogastrogram (EGG) electrodes to get myoelectrical readings
Diagnostic Test: MESG — MESG measures spatiotemporal properties of magnetic fields from the esophageal slow wave and allows characterization of the propagation of the slow wave in addition to evaluation of its frequency and power distribution
  Other Names: SQUID magnetometer
Diagnostic Test: High resolution manometry (HRM) — Dysphagia subjects will have undergone standard of care HRM to determine placement in the achalasia or hypercontractile/spastic disorder arms
  Arms: Achalasia subjects; Hypercontractile/spastic disorder subjects

SUMMARY:
The investigator proposes to study electrical activity reflective of esophageal motility in adults noninvasively by the use of multichannel electroesophagogram (EESG) and magnetoesophagogram (MESG) recordings.

DETAILED DESCRIPTION:
Dysphagia, or difficulty with swallowing, is a common symptom affecting nearly 9.4 million individuals or 4% of the US population. High resolution esophageal manometry is currently considered the gold standard test for evaluation and diagnosis of esophageal motility disorders, but given that it requires trans-nasal placement in a conscious patient, this test is highly uncomfortable and associated with significant patient dissatisfaction. There are currently no noninvasive tests or markers available to test esophageal function and motility.

In the upper gastrointestinal system, as in the heart, disruption of the electrical syncytium in disease produces measurable dysrhythmia. Recent modifications of the standard electrogastrogram (EGG) that have increased the number of leads to 25 (termed high-resolution EGG) have allowed enhanced spatio-temporal resolution of electric slow wave activity, and newer analytic techniques. Additionally, the magnetogastrogram (MGG) overcomes many of the inherent limitations of the standard EGG. The goal of this proposal is to harness similar technologies applied to the esophagus to develop high-resolution electroesophagogram (EESG) and magnetoesophagogram (MESG) as noninvasive clinical methods to quantify esophageal function and motility disorders, which could guide intervention for a large number of adult patients.

The main aims in this proposal are to develop a mathematical model of esophageal function and characterize phenotypes of esophageal motility disorders using EESG/MESG in healthy controls and esophageal dysmotility patients and determine how EESG/MESG rhythm and pattern abnormalities relate to physiologic function.

ELIGIBILITY:
Inclusion Criteria:

* Adults ≥ 18 years of age who are undergoing HRM for routine standard of care evaluation for esophageal motility.
* Normal control participants (ages ≥ 18 years) who have no known gastrointestinal complications.

Exclusion Criteria:

* Those with claustrophobia who cannot lie still under the SQUID for the length of time required
* Due to interference with signal acquisition, subjects with contraindication to undergoing an MRI scan as noted in the MRI Safety checklist by Vanderbilt University Medical Center (such as with heart pacemakers, metal implants, or metal chips or clips) will not undergo SQUID, but can still be eligible to do cutaneous EESG.
* Morbid obesity (these patients are potentially unable to lie under the current generation of SQUID devices)
* Patients with a history of cardiac arrhythmias or taking anticoagulants will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2019-09-04 (Actual); Primary Completion 2026-09 (Estimated); Study Completion 2026-09 (Estimated)

PRIMARY OUTCOMES:
Presence of diagnostic pattern | 3 months
  EESG and MESG wave patterns will be used to see if there is a diagnostic pattern that helps identify normal function vs. the motility disorders (achalasia or hypercontractile/spastic disorders)

CONTACTS AND LOCATIONS:
Overall Officials: Dhyanesh Patel, MD, Principal Investigator — Vanderbilt University Medical Center
Locations (1):
- Vanderbilt University Medical Center, Nashville, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
The investigators agree to the timely release and sharing of information to be no later than the acceptance for publication of the main findings from the final data set. Investigators are also committed to ensuring that all data are free of identifiers that would permit linkage to individual research participants as well as variables that could lead to deductive disclosure of the identity of individual subjects.
Time Frame: Immediately following publication. No end date.
Access Criteria: Investigators whose proposed use of the data has been approved by an independent review committee ("learned intermediary") identified for this purpose